CLINICAL TRIAL: NCT07347509
Title: An Investigation of the Acute Effects of BCAA, L-Arginine, and Placebo Supplementation on Anaerobic Performance, Speed, Agility, and Recovery in Elite Soccer Players
Brief Title: Acute Effects of BCAA and L-Arginine on Performance in Elite Soccer Players
Acronym: CST-SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gökhan Atasever, Associate Professor, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CST-SOCCER-2024; ID SBA-2025-15316 (Other Grant/Funding Number: Ataturk University BAP Project)
Record Dates: First submitted 2025-12-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ergogenic Support and Performance
Keywords: Football; BCAA; L-Arginine; Performance
MeSH Terms: interventions — Arginine; Amino Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- BCAA Supplementation Group (Experimental): Participants received a single acute oral dose of branched-chain amino acids (BCAA) prior to the anaerobic performance, speed, agility, and recovery tests.
  Interventions: Combination Product: BCAA
- L-Arginine Supplementation Group (Experimental): Participants received a single acute oral dose of L-arginine prior to the anaerobic performance, speed, agility, and recovery tests.
  Interventions: Dietary Supplement: L-Arginine
- MIX Supplementation Group (Experimental): Participants received a placebo supplement prior to the anaerobic performance, speed, agility, and recovery tests.
  Interventions: Dietary Supplement: bcaa and l arginine

INTERVENTIONS:
Combination Product: BCAA — A single acute oral dose of branched-chain amino acids (BCAA) administered prior to the anaerobic performance, speed, agility, and recovery tests.
  Arms: BCAA Supplementation Group
Dietary Supplement: L-Arginine — A single acute oral dose of L-arginine administered prior to testing.
  Arms: L-Arginine Supplementation Group
Dietary Supplement: bcaa and l arginine — A placebo supplement administered prior to testing.
  Arms: MIX Supplementation Group

SUMMARY:
his study aims to investigate the acute effects of a single pre-exercise dose of branched-chain amino acids (BCAA) and L-arginine supplementation on anaerobic performance, sprint speed, agility, lactate response, and post-exercise heart rate recovery in male football players competing in a youth development league.

Twenty-one football players participating in the T.F.F. U-19 Development League will be randomly assigned to one of three groups: BCAA (n = 7), L-arginine (n = 7), or placebo (n = 7). Participants will receive either 12 g of BCAA (4:1:1), 5 g of L-arginine, or an equivalent amount of maltodextrin, administered 1.5 hours before training.

Performance assessments will include 10 m and 20 m sprint tests, an agility test, the Wingate anaerobic power test, blood lactate measurements, and post-exercise heart rate recovery measurements taken at the 1st, 3rd, and 5th minutes of recovery.

Data will be analyzed using repeated measures analysis of variance to examine within- and between-group differences.Data obtained from the study were analyzed using the JASP 0.95.4 software. Pre-test and post-test values of the experimental and control groups were evaluated using Repeated Measures ANOVA. Effect size was determined using Eta Squared (η²), and differences between groups were identified using Tukey post hoc analysis. A 95% confidence interval was applied, and statistical significance was accepted at p < 0.05.

In the BCAA group, 20 m sprint performance (p < 0.05) and agility test results (p < 0.05) improved significantly compared to the control group. Additionally, heart rate recovery at the 3rd and 5th minutes was significantly faster in the BCAA group compared to both the L-arginine and placebo groups (p < 0.05). In the L-arginine group, no significant improvements were observed in sprint performance, agility, lactate response, or Wingate parameters compared to placebo. No significant differences were found between groups in lactate response or anaerobic power variables (peak, mean, and minimum power, and fatigue index) (p > 0.05).

A single dose of BCAA supplementation improves short-distance sprint performance, agility, and heart rate recovery in football players; however, it does not have a significant effect on anaerobic power or lactate response. Acute L-arginine supplementation did not produce a significant ergogenic effect on these parameters. The findings suggest that amino acid supplementation may produce more pronounced effects with chronic rather than acute application

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, placebo-controlled experimental trial to examine the acute effects of branched-chain amino acid (BCAA) and L-arginine supplementation on selected performance and physiological parameters in elite youth male football players.

A total of 21 male football players competing in the Turkish Football Federation (T.F.F.) U-19 Development League will be recruited for the study. Participants will be randomly allocated into three groups: BCAA supplementation group (n = 7), L-arginine supplementation group (n = 7), and placebo group (n = 7). Randomization will be performed using a computer-generated random allocation sequence. Both participants and investigators will be blinded to group assignments throughout the study.

Participants in the BCAA group will receive a single oral dose of 12 g BCAA in a 4:1:1 ratio, while the L-arginine group will receive 5 g of L-arginine. The placebo group will receive an equivalent amount of maltodextrin. All supplements will be administered 1.5 hours prior to the training session under standardized conditions.

Following supplementation, participants will complete a standardized warm-up protocol before undergoing performance assessments. Performance measures will include 10 m and 20 m sprint tests to assess sprint speed, an agility test to evaluate change-of-direction ability, and the Wingate anaerobic power test to assess anaerobic performance parameters. Blood lactate concentrations will be measured at specified time points, and heart rate recovery will be recorded at the 1st, 3rd, and 5th minutes following exercise.

All testing procedures will be conducted under similar environmental and training conditions to minimize external variability. Data collected from the assessments will be used to examine acute physiological and performance responses to the supplementation protocols using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

Male football players aged 19 years

Actively competing in a youth development or amateur football league

Minimum of 3 years of regular football training experience

Training at least 4 days per week

Free from musculoskeletal injury in the last 6 months

No use of nutritional supplements (including BCAA or L-arginine) for at least 4 weeks prior to the study

Voluntary participation with written informed consent

Exclusion Criteria:

Presence of any cardiovascular, metabolic, neurological, or chronic disease

Use of medications or supplements that may affect performance outcomes

History of surgery within the last 6 months

Known allergy or intolerance to BCAA or L-arginine

Smoking or alcohol abuse

Failure to comply with study protocol

Ages: 19 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Anaerobic Performance | Immediately after acute supplementation
  Anaerobic performance assessed using the Wingate Anaerobic Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)